CLINICAL TRIAL: NCT00947687
Title: A Randomized, Phase 1B, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Inhaled PUR003 on a Controlled Influenza Virus Challenge in Healthy Adult Subjects
Brief Title: Safety and Efficacy Study of Inhaled PUR003 on a Controlled Influenza Virus Challenge in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmatrix Inc. (Industry)
Collaborators: Retroscreen Virology Ltd. (Industry); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 601-0001P-00
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: influenza; healthy subject; virus inoculation; symptom scores; viral shedding; bioaerosol output
MeSH Terms: conditions — Influenza, Human | interventions — PUR003

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PUR003 (Experimental)
  Interventions: Drug: PUR003
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PUR003 — Twice-daily (BID) doses of PUR003 will be delivered via inhalation using a commercially available nebulizer for a total of 7 days
  Arms: PUR003
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objectives of the study are to demonstrate the effectiveness, safety and tolerability of multiple daily doses of inhaled PUR003, in comparison with placebo, in healthy adults experimentally inoculated with Influenza A/Wisconsin/67/2005 (H3N2) virus.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 45 years.
* In general good health determined by a screening evaluation ≤120 days prior to double-blind IMP administration and on the day of admittance to quarantine.
* Seronegative (NDA) for challenge virus.
* Have not been vaccinated for influenza virus since 2006 (as determined in the medical history) or had a known influenza infection in the current season, defined as in the last 12 months.

Exclusion Criteria:

* Presence or evidence of significant acute or chronic, uncontrolled medical or psychiatric illness.
* Abnormal pulmonary function as evidenced by clinically significant abnormality in spirometry.
* Health care workers (including doctors, nurses, medical students and allied healthcare professionals) anticipated to have patient contact within two weeks of discharge from quarantine.
* Intending to travel (to countries for which vaccinations are recommended or where high risk of infections exists).
* Presence of household member or close contact (until 14 days after discharge from quarantine) who is: less than 3 years of age; has any known immunodeficiency; is receiving immunosuppressant medications; is undergoing or soon to undergo cancer chemotherapy within 28 days of challenge.
* Subjects with diagnosed emphysema or chronic obstructive pulmonary disease (COPD); elderly residing in a nursing home, affected by severe lung disease or medical condition; or a transplant (bone marrow or solid organ) organ recipient
* Subjects with any history of asthma, COPD, pulmonary hypertension, reactive airway disease, or any chronic lung condition of any aetiology.
* Regular daily smokers during the 6 months prior to study entry or those who have a significant history of any tobacco use at any time (≥ total 10 pack year history = one pack a day for 10 years).
* Presence of any febrile illness or symptoms of upper or lower tract respiratory infection in the 28 days prior to viral inoculation (such subjects may be re-evaluated for enrolment after resolution of the illness).
* Receipt of any investigational drug within 3 months, or prior participation in a clinical trial of any influenza vaccine or medication within 1 year of participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of PUR003 as determined by incidence of adverse events (AEs); changes in physical examination, chest examination; pulmonary function; vital signs; electrocardiogram (ECG) and clinical laboratory assessments. | Day 6

SECONDARY OUTCOMES:
Subjected-reported symptom scores assessed both individually and as a composite score evaluating severity overall and at the time of peak symptom score | Day 6 of study
Quantitative viral shedding from nasal viral inoculation until day 6 | Day 0 to day 6
Change in bioaerosol output with treatment and after viral inoculation | Day -2 to day 6

CONTACTS AND LOCATIONS:
Overall Officials: John P Hanrahan, MD, Study Director — Pulmatrix Inc.
Locations (1):
- Guys Drug Research Unit (GDRU), Quintiles Ltd, London, United Kingdom